CLINICAL TRIAL: NCT04479930
Title: Development and Preliminary Evaluation of the Effects of an mHealth Web-Based Platform (HappyAir) on Adherence to a Maintenance Program After Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease: Randomized Controlled Trial
Brief Title: Effects of an mHealth Web-Based Platform (HappyAir) on Adherence to a Maintenance Program After Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Principal Investigator, bjreguera@ceu.es, Professor, CEU San Pablo University, CEU San Pablo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU017
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HappyAir Group (Experimental): The HappyAir app comprises two main parts: an educational program providing patients useful information and advice about their illness and data collection related to physical activity and disease.
  Interventions: Other: Pulmonary Care Web-Based App (HappyAir App)
- Control group (No Intervention): The control group only underwent the scheduled check-ups

INTERVENTIONS:
Other: Pulmonary Care Web-Based App (HappyAir App) — The HappyAir app reminded the HappyAir group daily to use the app, indicating that they record medication intake, daily exercise time (minutes), level of tiredness after the exercises (good, little tired, very tired, or exhausted), and daily mood (happy, little sad, sad, or very sad). The HappyAir integrated plan was designed as a model of a therapeutic program based on communication that introduced the figure of the therapeutic educator (physiotherapist or respiratory coach) in order to design interventions focused on the patients and their needs, with minimal intervention and presence, making the patients responsible for their self-care and management of their illness. Patient and educator shared responsibility.
  Arms: HappyAir Group

SUMMARY:
Objective: This study aimed to assess the effects of an integrated care plan based on an mHealth web-based platform (HappyAir) on adherence to a 1-year maintenance program applied after pulmonary rehabilitation in COPD patients.

Methods: COPD patients from three hospitals were randomized to a control group or an intervention group (HappyAir group). Patients from both groups received an 8-week program of pulmonary rehabilitation and educational sessions about their illness. After completion of the process, only the HappyAir group completed an integrated care plan for 10 months, supervised by an mHealth system and therapeutic educator. The control group only underwent the scheduled check-ups. Adherence to the program was rated using a respiratory physiotherapy adherence self-report (CAP FISIO) questionnaire. Other variables analyzed were adherence to physical activity (Morisky-Green Test), quality of life (Chronic Obstructive Pulmonary Disease Assessment Test, St. George's Respiratory Questionnaire, and EuroQOL-5D), exercise capacity (6-Minute Walk Test), and lung function.

ELIGIBILITY:
Inclusion Criteria:

* COPD patient.
* Aged between 55 and 85 years.
* Degree of severity II, III, or IV of the Global Initiative for Chronic Obstructive Lung Disease (GOLD) scale.
* Stable clinical situation (no exacerbations in the last 6 weeks).

Exclusion Criteria:

* Unstable cardiovascular disease or muscular, osteoarticular, auditory, visual, or central or peripheral nervous system impairment that prevents the performance of the rehabilitation program or evaluation tests.
* Cognitive impairment that makes it difficult to understand the education program and manage the HappyAir system

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Treatment Adherence | 10 months
  Adherence to the maintenance program was measured with the respiratory physiotherapy adherence self-report questionnaire (CAP PHYSIO).
  It consists of a total of 16 items, with a Likert scale to score each one, with 1 point as totally disagree and 4 points as totally agree. Three different dimensions of results are obtained: Total CAP, Perception and Adherence. The final rating scale is set to a range of minimum of 16 points (minimum adherence) to a maximum of 64 points (maximum adherence).

SECONDARY OUTCOMES:
Adherence to physical activity | 10 months
  Adherence to physical activity was measured with the therapeutic compliance questionnaire (Morisky-Green Test).
  It consists of a series of four contrast questions with a "yes/no" dichotomous answer, which reflects the patient's behavior with respect to compliance. It results in a score ranging from 0 (High adherence) to 4 (Low adherence).
Self-reported Quality of Life: EuroQOL-5D | 10 months
  Quality of life was measured with three different self-reported questionnaires, including the Chronic Obstructive Pulmonary Disease Assessment Test, St. George's Respiratory Questionnaire and EuroQOL-5D
Exercise Capacity | 10 months
  Exercise capacity was measured with the 6-Minute Walk Test (6MWT)

CONTACTS AND LOCATIONS:
Overall Officials: Begoña Jimenez Reguera, Msc, Principal Investigator — CEU San Pablo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez-Reguera B, Maroto Lopez E, Fitch S, Juarros L, Sanchez Cortes M, Rodriguez Hermosa JL, Calle Rubio M, Hernandez Criado MT, Lopez M, Angulo-Diaz-Parreno S, Martin-Pintado-Zugasti A, Vilaro J. Development and Preliminary Evaluation of the Effects of an mHealth Web-Based Platform (HappyAir) on Adherence to a Maintenance Program After Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jul 31;8(7):e18465. doi: 10.2196/18465. PMID 32513646